CLINICAL TRIAL: NCT06966570
Title: A Randomized, Single-Blind, Crossover Pilot Trial to Assess the Effects of Proprietary Beverages on Acute Appetite Hormone Response in Healthy Adults
Brief Title: Acute Appetite Hormone Response of Proprietary Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaklee Corporation (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry); Nlumn LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BIO-2503
Record Dates: First submitted 2025-04-29; First posted 2025-05-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: appetite, beverages, healthy adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Product A followed by Study Product B (Other)
  Interventions: Other: Study Product A: Mixed-macronutrient beverage; Other: Study Product B: Single-macronutrient beverage
- Study Product B followed by Study Product A (Other)
  Interventions: Other: Study Product A: Mixed-macronutrient beverage; Other: Study Product B: Single-macronutrient beverage

INTERVENTIONS:
Other: Study Product A: Mixed-macronutrient beverage — Participants will consume a beverage that contains mixed macronutrients.
Other: Study Product B: Single-macronutrient beverage — Participants will consume a beverage that contains a single macronutrient.

SUMMARY:
The primary objective of this study is to evaluate post-meal appetite hormones and appetite ratings, assessed using visual analog scale (VAS) questionnaires, in response to proprietary beverages in generally healthy adults.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate post-meal appetite hormones and appetite ratings, assessed using visual analog scale (VAS) questionnaires, in response to proprietary beverages in generally healthy adults compared to their baseline. It is hypothesized that beverages will result in an increase in appetite hormones and feelings of satiety compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ≥20 to ≤50 years of age.
2. BMI ≥18.5 and <25.0 kg/m2.
3. Self-reported regular consumer (≥5 days/week) of breakfast.
4. Women who are either pre- or post-menopausal. Premenopausal women that are not using hormonal contraceptives must have a history of regular menstrual cycles (21-35 d per cycle or at the investigator's discretion) for at least 3 months prior.
5. Willing to use personal smart phone and capable of downloading the Cronometer app for diet records.
6. Willing to adhere to all study procedures, including lifestyle considerations, and sign forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Is currently following, or planning to be on, a weight loss regimen at any time prior to or during the study.
2. Weight loss or gain >4.5 kg within 90 days.
3. History of gastrointestinal surgery for weight reducing purposes.
4. History of an eating disorder (e.g., anorexia nervosa or bulimia nervosa, binge eating) or extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan, vegetarian) at the discretion of the Clinical Investigator.
5. History of unconventional sleep patterns (e.g., night shift) or a diagnosed sleep disorder or chronic medical condition that may impact appetite (in the judgment of the Investigator).
6. Use of tobacco/nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months.
7. Use of hemp/marijuana products within 60 days. Occasional use (e.g., once or twice a month) within 60 days is allowed.
8. Unstable use of any prescription medication, where stable use is defined as no change in dose or medication type within 90 days.
9. Unstable use (initiation or change in dose) within 30 days of hormonal contraceptives.
10. Use of any dietary supplements, except for a conventional once daily multivitamin/mineral supplement.
11. Recent history of (within 12 months) or strong potential for alcohol or substance abuse.
12. Exposed to any non-registered drug product within 30 days prior.
13. A score of <7 on the Vein Access Scale Assessment.
14. History or presence, on the basis of the medical history or screening labs, of clinically important cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, gastrointestinal, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
15. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg).
16. Known allergy to any ingredients contained in the study product or study foods.
17. Any signs or symptoms of active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 days.
18. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
19. History of any major trauma or major surgical event within 2 months.
20. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential with unstable use (initiation or change in dose within 30 days) of sex hormones for contraception.
21. An employee or representative who has a financial interest in Shaklee Corporation.
22. Any condition the Investigator believes would interfere with the participant's ability to provide informed consent or comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) above baseline for appetite hormones | Up to 2 hours post-beverage consumption

SECONDARY OUTCOMES:
Positive area under the curve (AUC) for appetite hormones | Up to 2 hours post-beverage consumption
Time to Cmax (Tmax) for appetite hormones | Up to 2 hours post-beverage consumption
Individual and composite appetite visual analog scale (VAS) ratings | Up to 2 hours post-beverage consumption

CONTACTS AND LOCATIONS:
Overall Officials: Erin Barrett, PhD, Study Director — Shaklee Corporation
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No